CLINICAL TRIAL: NCT01974024
Title: Antiemetic Corticosteroid Rotation From Dexamethasone to Methylprednisolone to Prevent Dexamethasone-Induced Hiccup in Cancer Patients Treated With Chemotherapy: A Randomized, Single-Blind, Crossover Phase III Trial
Brief Title: Dexamethasone-induced Hiccup in Chemotherapy Patients Treated by Methylprednisolone Rotation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chung-Ang University (Other)
Collaborators: Gyeongsang National University Hospital (Other); Dong-A University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, In Gyu Hwang, In Gyu Hwang/Associate Professor, Chung-Ang University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GSNUH 2013-1
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Dexamethasone-induced Hiccup in Chemotherapy
Keywords: Dexamethasone; Hiccup; Chemotherapy; Methylprednisolone
MeSH Terms: conditions — Hiccup | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone (Experimental): Dexamethasone was replaced with methylprednisolone as an antiemetic.
  Interventions: Drug: methylprednisolone
- Dexamethasone (Active Comparator): Dexamethasone was re-administered in the cycle.
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — Adult patients who experienced DIH within 3 days after the administration of dexamethasone as an antiemetic were screened. Eligible patients were randomly assigned to receive dexamethasone or methylprednisolone as an antiemetic (randomization phase). In the next cycle of chemotherapy, the dexamethasone group received methylprednisolone and vice versa in the methylprednisolone group (crossover phase).
  Other Names: solu-medrol

SUMMARY:
The aims of this study were to investigate the feasibility of methylprednisolone rotation as treatment of DIH.

DETAILED DESCRIPTION:
we planned a randomized prospective trial for cancer patients with DIH. The objective of the present study was to determine whether the rotation of corticosteroids affects the incidence and intensity of DIH without compromising the antiemetic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* all solid cancer patients on chemotherapy
* age >18 years
* received dexamethasone as an antiemetic

Exclusion Criteria:

* brain metastases
* hiccups before dexamethasone administration
* uncontrolled diabetes mellitus
* uncontrolled esophagitis or peptic ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-31 (Actual)

PRIMARY OUTCOMES:
The intensities of hiccups | 2 months
  Clinically assessed every cycles(2-4weeks). The intensities of hiccups were assessed using a NRS.

SECONDARY OUTCOMES:
The intensities of emesis | 2 months
  CLinically assessed every cycles (2-4weeks) The intensities of emesis were assessed using a NRS.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hun Kang, M.D., Study Chair — Gyeongsang National University Hospital
Locations (2):
- South Korea (2):
  - Gyeongsang National University Hospital, Chiram-dong, Jinju-si, Gyeongsangnam-do
  - Chungang University Hospital, Dongjak-gu, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Go SI, Koo DH, Kim ST, Song HN, Kim RB, Jang JS, Oh SY, Lee KH, Lee SI, Kim SG, Park LC, Lee SC, Park BB, Ji JH, Yi SY, Lee YG, Yun J, Bruera E, Hwang IG, Kang JH. Antiemetic Corticosteroid Rotation from Dexamethasone to Methylprednisolone to Prevent Dexamethasone-Induced Hiccup in Cancer Patients Treated with Chemotherapy: A Randomized, Single-Blind, Crossover Phase III Trial. Oncologist. 2017 Nov;22(11):1354-1361. doi: 10.1634/theoncologist.2017-0129. Epub 2017 Jul 7. PMID 28687626